CLINICAL TRIAL: NCT01610479
Title: A Phase 1 Study of TAS-114 in Combination With S-1 in Patients With Advanced Solid Tumors
Brief Title: A Study of TAS-114 in Combination With S-1 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Taiho10050020
Record Dates: First submitted 2012-05-25; First posted 2012-06-04 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — TAS-114; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAS-114/S-1 (Experimental): TAS-114 plus S-1
  Interventions: Drug: TAS-114 + S-1

INTERVENTIONS:
Drug: TAS-114 + S-1

SUMMARY:
This is a phase 1 study of TAS-114 in combination with S-1 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase 1, open-label, non-randomized, dose-escalating safety, tolerability, and pharmacokinetic study of TAS-114 in combination with S-1 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 3 months
* Histological or cytological documentation of advanced solid tumors
* ECOG Performance Status of ≤ 1 (ECOG: Eastern Cooperative Oncology Group)
* Adequate bone marrow, liver and renal function
* Women of childbearing potential and men must agree to use adequate contraception

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of TAS-114 when used in combination with S-1 | 4 years

SECONDARY OUTCOMES:
Pharmacokinetic profiles (peak plasma concentration (Cmax) and area under the plasma concentration versus time curve (AUC) of TAS-114, S-1 components and its metabolite) | 4 years
Response rate | 4 years
Disease control rate | 4 years
Progression free survival | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Kashiwanoha, Kashiwa-shi, Chiba, Japan

REFERENCES:
- [Derived] Doi T, Yoh K, Shitara K, Takahashi H, Ueno M, Kobayashi S, Morimoto M, Okusaka T, Ueno H, Morizane C, Okano N, Nagashima F, Furuse J. First-in-human phase 1 study of novel dUTPase inhibitor TAS-114 in combination with S-1 in Japanese patients with advanced solid tumors. Invest New Drugs. 2019 Jun;37(3):507-518. doi: 10.1007/s10637-018-0697-3. Epub 2018 Dec 4. PMID 30511200